CLINICAL TRIAL: NCT02083770
Title: Randomized Controlled Clinical Trials Education Program for Hispanic Americans
Brief Title: Clinical Trials Education Program for Hispanic Americans
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: San Diego State University (Other)
Responsible Party: Principal Investigator, Georgia Robins Sadler, Professor, University of California, San Diego
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: CCT2525; NCI R25CA 130869 (Other: UCSD)
Record Dates: First submitted 2014-03-04; First posted 2014-03-11 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Cancer
Keywords: Hispanics; Patient Participation; Refusal to Participate; Education; Clinical Trials
MeSH Terms: conditions — Neoplasms; Patient Participation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cancer Clinical Trials Education Program (Experimental): Cancer Clinical Trials Education Program is offered to English- and Spanish-speaking Hispanics in the experimental arm. This program was designed to promote increased clinical trials literacy among Hispanic Americans. Increased clinical trials knowledge and a better understanding of clinical trials is anticipated to create more positive attitudes, and perceptions about clinical trials among Hispanic Americans.
  Interventions: Behavioral: Cancer Clinical Trials Education Program
- Neighborhood Watch Education Program (Placebo Comparator): The Neighborhood Watch Program created by the Bureau of Justice Assistance and the National Crime Prevention Council was selected for inclusion in the control arm of this study. It provided participants with a program of equivalent length and format, as well as an equivalent focus on improving the well-being of Hispanic Americans. It also provided an opportunity to evaluate the impact of the Neighborhood Watch Program.
  Interventions: Behavioral: Cancer Clinical Trials Education Program

INTERVENTIONS:
Behavioral: Cancer Clinical Trials Education Program — Hispanic Americans are underrepresented in cancer clinical trials. The purpose of this study is to develop and test programs designed to reduce barriers and increase facilitators associated with cancer clinical trials participation for Hispanic Americans.

SUMMARY:
Hispanic Americans are underrepresented in cancer clinical trials. The purpose of this study is to develop and test programs designed to reduce barriers and increase facilitators associated with cancer clinical trials participation for Hispanic Americans.

DETAILED DESCRIPTION:
Hispanic Americans are underrepresented in cancer clinical trials. The purpose of this study is to develop and test education programs designed to reduce barriers and Increase facilitators associated with cancer clinical trials participation for Hispanic Americans. Focus groups were conducted with Hispanic American men and women to obtain culturally-linked attitudes related to clinical trials participation. This information was used to create a prototypic educational program anticipated to increase participation in clinical trials. It was then vetted and honed via additional focus groups.

Simultaneously, a validation study was conducted with Hispanic Americans for a packet of psychosocial instruments that could be used for a subsequent randomized controlled trial to evaluate the impact of the clinical trials education program.

The finalized clinical trials education program was tested via a randomized controlled trial. Participants assigned to the experimental group received the clinical trials education program, while participants in the control arm were administered a comparable, but non-relevant education program. Recruitment to this study has been completed.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified as Hispanic American
* At least 21 years of age
* Sufficiently literate to comprehend written and spoken testing materials in English or Spanish
* Living in southern California
* Mentally competent to complete the informed consenting process

Exclusion Criteria:

-

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1034 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Change in Participants' Clinical Trials-Related Knowledge, Attitudes and Beliefs From Baseline to First Follow-up | Change from baseline to first follow-up (immediately after receiving intervention)
  To assess the impact of the intervention arm on participants' knowledge, attitudes, and perceptions related to clinical trials, they were asked to complete the same surveys given at baseline during post-intervention immediately after intervention.
Change in Participants' Clinical Trials-Related Knowledge, Attitudes and Beliefs From Baseline to Second Follow-up | Change from baseline to second follow-up (three months after receiving intervention)
  At the three-month follow-up, participants were mailed the final packet of survey instruments to complete and return in a stamped, self-addressed envelope.

SECONDARY OUTCOMES:
Willingness to Participate in Research | Two weeks after receiving intervention
  Two weeks after receiving the intervention, participants were mailed an invitation to participate in a different research study by a researcher not previously known to them, to assess whether the intervention influenced behavior related to clinical trials invitations.

CONTACTS AND LOCATIONS:
Overall Officials: Georgia R Sadler, PhD, Principal Investigator — UC San Diego Moores Cancer Center; Vanessa L Malcarne, PhD, Principal Investigator — San Diego State University
Locations (1):
- UC San Diego Moores Cancer Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Merz EL, Malcarne VL, Roesch SC, Riley N, Sadler GR. A multigroup confirmatory factor analysis of the Patient Health Questionnaire-9 among English- and Spanish-speaking Latinas. Cultur Divers Ethnic Minor Psychol. 2011 Jul;17(3):309-316. doi: 10.1037/a0023883. PMID 21787063